CLINICAL TRIAL: NCT02087527
Title: Use of Corticosteroids in Children Hospitalized With Cellulitis: Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Use of Corticosteroids in Children With Cellulitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Calculated sample size not achieved
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HGNPE-128-2013
Record Dates: First submitted 2014-02-19; First posted 2014-03-14 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Cellulitis
Keywords: Cellulitis; Soft Tissue Infections; Skin Diseases, Infectious; Corticosteroids; Glucocorticoids; Dexamethasone
MeSH Terms: conditions — Cellulitis; Soft Tissue Infections; Skin Diseases, Infectious | interventions — Dexamethasone; Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CORTICOSTEROID (Experimental): In addition to standard care for cellulitis, subject will receive intravenous Dexamethasone (8mg/2ml) 0.15 mg/kg/dose every 6 hours for the first 48 hours
  Interventions: Drug: Dexamethasone
- NORMAL SALINE (Placebo Comparator): In addition to standard care for cellulitis, subject will receive normal saline solution administered intravenously using the same volume as the active drug group every 6 hours for the first 48 hours
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexamethasone — IV Dexamethasone 0.15 mg/kg every 6 hours for 48 hours
  Other Names: Decadron
  Arms: CORTICOSTEROID
Drug: Normal Saline — IV normal saline every 6 hours for 48 hours
  Other Names: ClNa 0.9%
  Arms: NORMAL SALINE

SUMMARY:
The aim of this study is to evaluate the efficacy of addition of corticosteroid therapy to antibiotic treatment during the first 48 hours of admission to the hospital in patients with cellulitis and its impact in the duration of the stay.

DETAILED DESCRIPTION:
Cellulitis is a common skin and soft tissue infection in the pediatric population.

Although most of the time treatment could be administered on an ambulatory setting , sometimes it may require hospitalization and parenteral antibiotic administration. Using corticosteroids during antibiotic treatment may reduce inflammation and length of stay.

Objective: to evaluate the efficacy of using corticosteroids as adjuvant treatment during the first 48 hours of treatment after hospitalization in patients with cellulitis.

Patients and methods: this is a double blind, randomized, controlled trial that will take place at pediatric hospital, during one year. It will include children aged 1 month to 18 years, admitted due to cellulitis. Once included in the clinical trial, the patients will be randomized to receive dexamethasone 0,6 mg/kg/day or placebo (saline solution) during the first 48 hours. Considering an average stay of 4 ± 2 days, we calculated a sample size of 124 children (62 children per group) to detect a 25% difference (1 day reduction) in the length of stay, with a power of 80% and a confidence of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Children Aged 1 month to 18 years
* Hospitalized due to cellulitis
* Patients who have given their written informed consent to participate

Exclusion Criteria:

* Skin chronic diseases
* Immunodeficiency (primary or acquired)
* Chronic use of systemic corticosteroids
* Sepsis
* Varicella
* History of adrenal insufficiency
* Pregnancy or breast feeding
* Uncontrolled diabetes mellitus
* Known hypersensitivity to systemic or topical corticosteroids
* Patient undergoing immunosuppressive therapy for another disease
* Participation in another drug biomedical research
* Any other contraindication for treatment with corticosteroids

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Length of stay | participants will be followed for the duration of hospital stay, an expected average of 5 days

SECONDARY OUTCOMES:
Fever duration | participants will be followed for the duration of hospital stay, an expected average of 5 days
Change in erythema size | Measured at admission and after 48 hours (at the end of corticosteroids treatment)
Need to change antibiotic treatment | participants will be followed for the duration of hospital stay, an expected average of 5 days
Abscessation or spontaneous drainage | participants will be followed for the duration of hospital stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano G Gigliotti, MD, Study Director — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de NIños Pedro de Elizalde, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bergkvist PI, Sjobeck K. Antibiotic and prednisolone therapy of erysipelas: a randomized, double blind, placebo-controlled study. Scand J Infect Dis. 1997;29(4):377-82. doi: 10.3109/00365549709011834. PMID 9360253
- [Background] McGowan JE Jr, Chesney PJ, Crossley KB, LaForce FM. Guidelines for the use of systemic glucocorticosteroids in the management of selected infections. Working Group on Steroid Use, Antimicrobial Agents Committee, Infectious Diseases Society of America. J Infect Dis. 1992 Jan;165(1):1-13. doi: 10.1093/infdis/165.1.1. No abstract available. PMID 1727879
- [Background] Thompson J. Role of glucocorticosteroids in the treatment of infectious diseases. Eur J Clin Microbiol Infect Dis. 1993;12 Suppl 1:S68-72. doi: 10.1007/BF02389882. PMID 8477768
- [Background] Fritz KA, Weston WL. Systemic glucocorticosteroid therapy of skin disease in children. Pediatr Dermatol. 1984 Jan;1(3):236-45. doi: 10.1111/j.1525-1470.1984.tb01123.x. PMID 6387668
- [Background] Jaussaud R, Kaeppler E, Strady C, Beguinot I, Waldner A, Remy G. [Should NSAID/corticoids be considered when treating erysipelas?]. Ann Dermatol Venereol. 2001 Mar;128(3 Pt 2):348-51. French. PMID 11319363
- [Background] Kilburn SA, Featherstone P, Higgins B, Brindle R. Interventions for cellulitis and erysipelas. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD004299. doi: 10.1002/14651858.CD004299.pub2. PMID 20556757
- [Background] Pushker N, Tejwani LK, Bajaj MS, Khurana S, Velpandian T, Chandra M. Role of oral corticosteroids in orbital cellulitis. Am J Ophthalmol. 2013 Jul;156(1):178-183.e1. doi: 10.1016/j.ajo.2013.01.031. Epub 2013 Apr 24. PMID 23622565
- [Derived] Kornelsen E, Mahant S, Parkin P, Ren LY, Reginald YA, Shah SS, Gill PJ. Corticosteroids for periorbital and orbital cellulitis. Cochrane Database Syst Rev. 2021 Apr 28;4(4):CD013535. doi: 10.1002/14651858.CD013535.pub2. PMID 33908631